CLINICAL TRIAL: NCT00311389
Title: A 12-Month Study to Evaluate the Efficacy and Safety of Once-Daily Instillation of Combination Glaucoma Therapy in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-28
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Glaucoma, Open-angle; Ocular Hypertension
Keywords: Glaucoma; POAG; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — Travoprost; Timolol; Ophthalmic Solutions; Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Travoprost/Timolol (Experimental): 1 drop in the affected eye(s) once daily in the morning for 12 months
  Interventions: Drug: Travoprost 0.004%/Timolol maleate 0.5% ophthalmic solution
- Latanoprost/Timolol (Active Comparator): 1 drop in the affected eye(s) once daily in the morning for 12 months
  Interventions: Drug: Latanoprost 0.005%/Timolol 0.005% ophthalmic solution

INTERVENTIONS:
Drug: Travoprost 0.004%/Timolol maleate 0.5% ophthalmic solution — Investigational ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: Travoprost/Timolol
Drug: Latanoprost 0.005%/Timolol 0.005% ophthalmic solution — Commercially marketed ophthalmic solution intended for the treatment of open-angle glaucoma or ocular hypertension
  Arms: Latanoprost/Timolol

SUMMARY:
The purpose of this study is to evaluate the intraocular pressure(IOP)-lowering efficacy of a combination IOP-lowering therapy in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

- As specified in protocol

Exclusion Criteria:

- As specified in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2003-01; Primary Completion 2004-09 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Mean Intraocular Pressure (IOP) | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- European Facilitiies, Puurs, Belgium